CLINICAL TRIAL: NCT01575353
Title: Nasal High-flow Oxygen Therapy vs Standard Oxygen Therapy Via Venturi Mask in the Post-extubation Period
Brief Title: Nasal High-flow Versus Venturi Mask Oxygen Therapy in the Post-extubation Period
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Salvatore Maurizio MAGGIORE, Assistant Professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1399/10
Record Dates: First submitted 2010-12-13; First posted 2012-04-11 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Venturi mask (Active Comparator): After extubation, patients will receive oxygen therapy through the standard Venturi mask (control)
  Interventions: Device: Venturi mask
- Nasal high-flow (Active Comparator): After extubation, patients will receive oxygen therapy through the nasal high-flow (intervention)
  Interventions: Device: Nasal high-flow

INTERVENTIONS:
Device: Venturi mask — The patients will receive oxygen delivered through a conventional Venturi mask. The FiO2 (color coded) will be adjusted in order to obtain a SpO2 between 92% and 98% in hypoxemic patients and between 88% and 95% in hypercapnic patients.
  Arms: Venturi mask
Device: Nasal high-flow — The patients will receive oxygen delivered through the nasal high-flow system (Optiflow™). The FiO2 will be adjusted in order to obtain a SpO2 between 92% and 98% in hypoxemic patients and between 88% and 95% in hypercapnic patients. Gas flow will be set at 50l/min.
  Other Names: Optiflow™
  Arms: Nasal high-flow

SUMMARY:
The aim of the study is to compare two devices for oxygen therapy, nasal high-flow and Venturi mask, in critically ill patients in the post-extubation period. The hypothesis is that nasal high-flow may be superior to the Venturi mask in terms of oxygenation

DETAILED DESCRIPTION:
Acute respiratory failure is one the most common reason for admission and mechanical ventilation is the most frequent procedure performed in the intensive care unit (ICU). After extubation, oxygen therapy is commonly used to correct residual impairment in oxygenation. Oxygen therapy is usually performed via a Venturi mask allowing to deliver predetermined oxygen concentrations. The face mask is used in the place of nasal cannula in part because patients with acute respiratory failure (ARF) breath preferentially through an open mouth rather than the nose. The mask may, however, reduce comfort and patients with ARF, who are often agitated and poorly cooperative, may displace or self-remove the mask. Given that oxygen delivered to the patient is dry, clinical practice guidelines recommend humidifying the oxygen when above 4 l/min in the ICU setting, because the humidification function of the nasal mucosa can be insufficient at high oxygen flow rates and/or the critically ill patient with ARF often breathes through the mouth. Breathing dry oxygen could provoke dryness of the mouth, nose, throat and respiratory tract, resulting in discomfort and pain that are frequent in the ICU setting. Breathing dry air by the nose may also lead to the alteration of the mucociliary transport system and cause an increase of airway resistance in healthy subjects. However, there are no recommendations concerning the type of humidification device to use.

High-flow oxygen therapy is commonly practiced in the ICU. Recently, a method was described in which high-flow oxygen is delivered through a nasal cannula with an active humidification system that optimizes oxygen administration in patients with ARF (Optiflow, Fisher & Paykel, New Zealand). This system has several theoretical advantages. The delivery of high flows decreases dilution of the inhaled oxygen and, by matching patient's peak flow, allows accurate delivery of the set FiO2 throughout the whole inspiratory phase. In addition, a flow-dependent effect of continuous positive airway pressure, possibly due to an air entrainment mechanism, has been documented in healthy volunteers and in patients with COPD. Lastly, the use of high humidity levels may prevent damage to the ciliated epithelium of the airways, maintain mucociliary system activity, and facilitate the elimination of secretions. Through these effects, this new device for high-flow oxygen therapy has the potential to be effective and to improve tolerance to the treatment more than conventional systems for oxygen therapy, such as the Venturi mask.

In the present randomized, controlled trial, the investigators will compare two devices for oxygen therapy, nasal high-flow oxygen therapy and the standard Venturi mask, in critically ill patients who need oxygen in the post-extubation period. The hypothesis is that nasal high-flow is superior to the Venturi mask in terms of oxygenation

ELIGIBILITY:
Inclusion Criteria:

* Mechanical ventilation > 24h
* Successful spontaneous breathing trial conducted for a period of 30-120 min.
* PaO2/FiO2 ≤ 300 at the end of the spontaneous breathing trial preceding extubation

Exclusion Criteria:

* age<18 years
* pregnancy
* tracheostomy
* need of NIV post-extubation (prophylactic NIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-12; Primary Completion 2011-05 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Oxygenation (PaO2/FiO2 ratio) | Up to 48 hours after extubation
  Arterial blood gases will be collected and the PaO2/FiO2 ratio will be measured 1, 3, 6, 12, 24, 36 and 48 hours after enrollment.

SECONDARY OUTCOMES:
Patient's discomfort, need for non-invasive ventilation, endotracheal intubation, oxygen desaturations, interface displacements | 48 hours after enrollment
  Patient's discomfort, the need and causes for non-invasive ventilation or endotracheal intubation, episodes of oxygen desaturation (defined as SpO2 < 92% or < 88% in hypercapnic patients with chronic obstructive pulmonary disease) and episodes of displacement of the device for oxygen delivery (as estimated by nurses) will be recorded in the 48h study period. Patient's discomfort related to the device used for oxygen therapy and related to the degree of humidification will be assessed by using a numerical rating scale from 0 (no discomfort) to 10 (maximum imaginable discomfort). Patients will be asked to rate their discomfort with the used device and discomfort symptoms will be determined for the dryness of the delivered oxygen (dryness of the mouth, throat, nose, difficulty to swallow and throat pain).

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Maurizio Maggiore, MD, PhD, Principal Investigator — Catholic University of the Sacred Heart; Massimo Antonelli, MD, Study Director — Catholic University of the Sacred Heart
Locations (2):
- Italy (2):
  - ICU, "Maggiore della Carità", University Hospital, Novara, Novara
  - ICU "A. Gemelli" University Hospital, Rome, Rome

REFERENCES:
- [Derived] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980